CLINICAL TRIAL: NCT06923033
Title: Aim 1: Augmented Reality as an Adjunct to Quitline Counseling for Smoking Cessation
Brief Title: Aim 1: App for Reducing Cravings to Smoke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MCC-21980 Aim1; R01DA055298 (NIH)
Record Dates: First submitted 2025-04-09; First posted 2025-04-11 (Actual); Results first posted 2025-06-15 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aim 1: Update an existing smartphone App (Experimental): An existing study app will be updated to be engaging, user-friendly treatment tool, and verify user satisfaction.
  Interventions: Behavioral: Smartphone App

INTERVENTIONS:
Behavioral: Smartphone App — Participants will download a study app that will allow them to track smoking urges and abstinence. Access to augmented reality will become available after 48 hours of self-reported abstinence.

SUMMARY:
The aim of this study is to update a recently developed study-related smartphone application to reduce cravings to smoke to be an engaging, user-friendly treatment tool, and verify user satisfaction

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* Daily smokers that have quit smoking within the past 3 months (Aim 1) or currently smoking ≥ 3 cigarettes per day for the past year (Aim 2)
* Functioning telephone number
* Owns a smart phone capable of supporting AR and willing to download the app
* Can speak, read and write in English

Exclusion Criteria:

* Has another household member already enrolled in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2023-10-09 (Actual); Primary Completion 2023-11-02 (Actual); Study Completion 2023-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Vinci, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aim 1: Update an Existing Smartphone App
Started | 14
Completed | 10
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Aim 1: Update an Existing Smartphone App
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.9 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: System Usability Scale (Aim 1)
Description: Participants' perception of usability and learnability of the app will be measured using 10 items on a 5-point Likert scale. Scores range from 0 to 100, with higher scores indicating better usability.
Time Frame: At 1 week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aim 1: Update an Existing Smartphone App
Number analyzed (Participants) | 10
score on a scale | 70.3 (20.1)

2. Secondary Outcome: User Satisfaction (Aim 1)
Description: One Likert scale item will capture participants' satisfaction with the app. The Likert scale is from 1 to 4, with higher score indicating greater satisfaction.
Time Frame: At 1 week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aim 1: Update an Existing Smartphone App
Number analyzed (Participants) | 10
score on a scale | 3.4 (0.6)

ADVERSE EVENTS:
Description: Death, serious adverse events, and other (non-serious adverse events) were not assessed for the study.
Arm/Group | Aim 1: Update an Existing Smartphone App
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-02-06): https://cdn.clinicaltrials.gov/large-docs/33/NCT06923033/Prot_SAP_000.pdf